CLINICAL TRIAL: NCT00154271
Title: Effects of Blood Pressure Reduction on High Sensitivity C-Reactive Protein (hsCRP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAH631DUS02
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-08

CONDITIONS: Hypertension
Keywords: Hypertension (HTN); High Sensitivity C-Reactive Protein
MeSH Terms: conditions — Hypertension | interventions — Valsartan

INTERVENTIONS:
Drug: Valsartan, Valsartan HCT

SUMMARY:
The study compares the efficacy of an aggressive versus a moderate initial antihypertensive regimen to reduce blood pressure in patients with Stage 2 hypertension. Additionally, the study examines the effects of blood pressure reduction on the levels of high sensitivity hsCRP. Although the main goal is to determine the overall effect of blood pressure reduction on hsCRP levels, analysis will also evaluate whether an aggressive antihypertensive regimen is more effective than a moderate one in reducing hsCRP levels.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 2 hypertension as defined by the mean of three (3) repeated seated BP measurements of: SBP of 160 to 185 mmHg, inclusive and/or DBP of 100 to 109 mmHg, inclusive.
2. Patients must have documentation of serum creatinine equal or <2.0 mg/dL, serum potassium equal or >3.5 and equal or <5.5 mmol/L, and serum AST or ALT <2xULN obtained within 3 months prior to Visit 1.
3. Patients must have documentation of HbA1C equal or <11.0 % obtained within 1 month prior to Visit 1.

Exclusion Criteria:

1. History of secondary hypertension.
2. Pharmacologic antihypertensive therapy with ACE inhibitors, angiotensin receptor blockers, or aldosterone blockers within 3 months prior to Visit 1, or with thiazide diuretics within 1 month prior to Visit 1. The use of other classes of agents which lower BP but are being used for other therapy or for HTN, are allowed as long as these agents are started at least 3 months prior to randomization, are not initiated after enrollment and doses remain unchanged during the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1677 (Actual)
Dates: Start 2004-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 6 in mean sitting blood pressure (SD)
Change from baseline to Week 12 in median plasma hsCRP
Change from baseline to Week 6 in median plasma hsCRP

SECONDARY OUTCOMES:
Proportion of responders with change in systolic BP
Time to first SBP reduction
Proportion of subjects achieving SBP control
Change in mean sitting DBP
Change in hsCRP for subjects with baseline hsCRP greater or equal to 3.0 mg/L

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

REFERENCES:
- [Derived] Everett BM, Glynn RJ, Danielson E, Ridker PM; Val-MARC Investigators. Combination therapy versus monotherapy as initial treatment for stage 2 hypertension: a prespecified subgroup analysis of a community-based, randomized, open-label trial. Clin Ther. 2008 Apr;30(4):661-72. doi: 10.1016/j.clinthera.2008.04.013. PMID 18498915